CLINICAL TRIAL: NCT03284190
Title: Scandinavian Multicentre Acute Subdural Hematoma (SMASH) Study: A Multi-national Population-based Consecutive Cohort
Brief Title: Scandinavian Multicentre Acute Subdural Hematoma (SMASH) Study
Acronym: SMASH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Jiri Bartek, MD, Karolinska University Hospital
Other Study IDs: SMASH
Record Dates: First submitted 2017-03-14; First posted 2017-09-15 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Acute Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural, Acute | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- ASDH Copenhagen, Denmark
  Interventions: Procedure: Surgery
- ASDH Odense, Denmark
  Interventions: Procedure: Surgery
- ASDH Århus, Denmark
  Interventions: Procedure: Surgery
- ASDH Ålborg, Denmark
  Interventions: Procedure: Surgery
- ASDH Lund, Sweden
  Interventions: Procedure: Surgery
- ASDH Linköping, Sweden
  Interventions: Procedure: Surgery
- ASDH Gothenburg, Sweden
  Interventions: Procedure: Surgery
- ASDH Stockholm, Sweden
  Interventions: Procedure: Surgery
- ASDH Uppsala, Sweden
  Interventions: Procedure: Surgery
- ASDH Umeå, Sweden
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Surgery

SUMMARY:
In a multi-national population-based cohort, the investigators want to compare the clinical course and clinical outcome of elderly patients (≥70 y/o) compared with younger patients (< 70 y/o) with acute subdural hematoma treated surgically. An improved understanding of the clinical outcome and the prognostic factors of acute subdural hematomas would allow physicians to make better decisions about treatment options in traumatic ASDH in the elderly population.

DETAILED DESCRIPTION:
Primary endpoint:

In a population based study to evaluate 30-day mortality (perioperative death) in younger versus elderly (≥70 years) patients with ASDH.

Secondary endpoint(s):

1. Describe pattern of care in younger versus the elderly
2. Clinical outcome (Glasgow outcome scale at 6-months (range, 3-12) follow-up in younger versus elderly (≥70 years) patients with ASDH:

   * Good outcome predefined as GOS 4-5
   * Unfavourable outcome predefined as GOS 1-3
3. 30-day morbidity (according to the Ibanez classification) in younger versus elderly (≥70 years) patients with ASDH.
4. To assess the effect of age as an independent prognostic factor in traumatic ASDH for outcome (GOS) in the elderly (≥70 years) using a three-step approach

   1. Match elderly (cases) with younger (controls) patients with respect to

      1. GCS at admission to treating hospital according to severity - mild (GCS 14-15), moderate (GCS 9-13), severe (GCS 3-8)
      2. Midline-shift (with a cut off of > 10 mm)
      3. Dilated pupil(s) (yes/no)
   2. Using a multivariable approach with all patients including age (continuous model) to identify independent predictors of an unfavourable outcome (GOS 1-3)
   3. Using a multivariable approach including age as a continuous variable within the elderly population (≥70 years) to identify independent predictors of an unfavourable outcome among the oldest (GOS 1-3)

ELIGIBILITY:
Inclusion Criteria:

* Surgically treated ASDH patients

Exclusion Criteria:

* Post-operative ASDH (i.e. inclusion criteria post-traumatic)
* Intracranial surgery within 6 months prior to trauma
* Permanent intracranial device (i.e DBS electode, VP shunt etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Surgically treated patients with acute subdural hematoma
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2018-03-06 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
30-day mortality (yes vs. no) in younger versus elderly | 30-day mortality after surgery
  30-day mortality (yes vs. no) in younger versus elderly

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bartek J Jr, Laugesen C, Mirza S, Forsse A, Petersen MA, Corell A, Dyhrfort PW, Redebrandt HN, Reen L, Zolfaghari S, Tobieson L, Carlsvard B, Bergholt B, Bashir A, Soerensen P, Bilgin A, Johansson C, Lindvall P, Forander P, Bellander BM, Springborg JB, Jakola AS. Scandinavian Multicenter Acute Subdural Hematoma (SMASH) Study: Study Protocol for a Multinational Population-Based Consecutive Cohort. Neurosurgery. 2019 Mar 1;84(3):799-803. doi: 10.1093/neuros/nyy173. PMID 29762769